CLINICAL TRIAL: NCT02876445
Title: Assessment Study on Family Burden in Overall Care of Patient With Huntington Disease
Brief Title: Caregiver Burden in Huntington's Disease
Acronym: PHRI-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NI10059
Record Dates: First submitted 2016-07-31; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-07

CONDITIONS: Caregiver of Huntington's Disease Patient
Keywords: Huntington's disease; Caregiver; ZARIT burden scale
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caregiver Evaluation (Other): ZARIT Burden Interview
  Interventions: Other: ZARIT Burden Interview

INTERVENTIONS:
Other: ZARIT Burden Interview — ZARIT Burden Interview completed Day 0 and 1 year

SUMMARY:
Huntington's disease (HD) is a rare inherited neurodegenerative disorder, progressing between 15 and 20 years and affecting one person out of 10.000. In France, it concerns some 6.000 patients symptomatic and 12 000 asymptomatic carriers.

Few extensive researches have been conducted on the progression of the disease, which is defined in the literature in 5 stages in a functional approach.

Therapeutically, no cure for HD is currently validated but only symptomatic treatments. There's various treatment options: medicated, humans (physiotherapy, speech therapist, occupational therapist, ..).

Although these treatment options do not prevent the progression of the disease, their combination associated with a stimulating environment may slow the decline of physical, intellectual and psychic abilities of patients.

In social terms, patients with HD require sustained support, especially in cases of family isolation.

The behavioural, gaiting and eating disorder as well as the communications difficulties make it difficult support daily for the entourage. The caregivers are sometimes dealing with untenable situations. Home care services, which are crucial to alleviating dependency, relieve family caregivers but are for the most severe patient.

Moreover, the justified placement decision in an institution generates a feeling of guilt for the family.

The caregiver is the person who brings non-professional assistance , partly or wholly , to a dependent member of his entourage , for the activities of daily living. This regular care may be provided permanently or not. It can take many forms, such as , care , nursing , support to education and social life , administrative procedures , psychological support .

Caregivers have their lives profoundly reshaped. They are often forced to give up some of their habits , give up their future plans , change their relationships. The commitment of caregivers with patients with Huntington's disease actually sounds on their mental and physical health, as well as their social and professional life

Very few studies have been conducted to measure the difficulties and implications of these caregivers.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18
* Primary caregiver of patient with Huntington's disease
* Non- institutionalized Patient
* stage 1-4 (no institutionalization within 2 years)
* written consent

Exclusion Criteria

- Not agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluation with ZARIT's scale of the burden level of the management of a patient with Huntington's disease by his caregiver | 1 year

SECONDARY OUTCOMES:
Measuring social impact of the disease using the under score of ZARIT's scale for the patient and the caregiver | 1 year
Measuring professional impact of of the disease using the under score of ZARIT's scale for the patient and the caregiver | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure BOURHIS, Senior Health Manager, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Youssov K, Audureau E, Vandendriessche H, Morgado G, Layese R, Goizet C, Verny C, Bourhis ML, Bachoud-Levi AC. The burden of Huntington's disease: A prospective longitudinal study of patient/caregiver pairs. Parkinsonism Relat Disord. 2022 Oct;103:77-84. doi: 10.1016/j.parkreldis.2022.08.023. Epub 2022 Aug 24. PMID 36084356